CLINICAL TRIAL: NCT02229500
Title: Regulating Appetite by Targeting Nutrient Delivery in the Gut
Brief Title: Investigating Optimal Propionate Delivery to the Colon Using Stable Isotope Labeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scottish Universities Environmental Research Centre (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BB/L004259/1_SUERC_1
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Optimum Propionate Delivery to the Large Intestine
Keywords: Propionate; Microbiome; Dietary Fibre; Short chain fatty acids
MeSH Terms: interventions — Inulin; Propionates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Inulin control, 10g/d for 7 days. Isotope and appetite measurements on day 7
  Interventions: Dietary Supplement: Inulin
- Delivery system 1 (Experimental): Delivery system, 28.5% w/w propionate, 10g/d for 7 days. Isotope and appetite measurements on day 7.
  Interventions: Dietary Supplement: 2.5 g of propionate
- Delivery system 2 (Experimental): Delivery system, 54% w/w propionate, 10g/d for 7 days. Isotope and appetite measurements on day 7.
  Interventions: Dietary Supplement: 5 g of propionate

INTERVENTIONS:
Dietary Supplement: Inulin
  Other Names: Beneo-Orafti HP
  Arms: Control
Dietary Supplement: 2.5 g of propionate — This system delivers approximately 2.5 g of propionate to the colon in a 10g dose.
  Arms: Delivery system 1
Dietary Supplement: 5 g of propionate — This delivers approximately 5g of propionate to the colon per 10g dose
  Arms: Delivery system 2

SUMMARY:
Obesity, with its associated co-morbidities, is a major public health challenge. It is estimated that by 2050, 60% of men and 50% of women will be clinically obese. Obesity is associated with increased risk of developing diabetes, cardiovascular disease, and certain cancers. The increasing epidemic of obesity has necessitated the study of the complex mechanisms underlying energy homeostasis. Food intake, energy balance and body weight are tightly regulated by the hypothalamus, brainstem and reward circuits, on the basis both of cognitive inputs and of diverse humoral and neuronal signals of nutritional status. Several gut hormones, including glucagon-like peptide-1 (GLP-1) and peptide YY3-36 (PYY), have been shown to play an important role in regulating short-term food intake. Peripheral administration of PYY or GLP-1 enhances satiety and reduces food intake in animals and man. PYY, GLP-1 along with a host of other hormones are produced by the gut in response to nutrient availability in different regions of the gut and provide an exquisite mechanism of nutrient sensing in response to dietary intake. These hormones therefore represent potential targets in the development of novel anti-obesity treatments. A novel and attractive strategy to induce appetite regulation is the enrichment of foods with components that stimulate the release of GLP-1 and PYY. The short chain fatty acids (SCFA) produced by microbial fermentation of dietary fibre in the colon have been shown to stimulate the release of PYY and GLP-1 from rodent enteroendocrine L cells, via stimulation of the G-protein coupled free fatty acid receptors (FFAR) on colonic L cells. Of the SCFAs produced by colonic fermentation of dietary fibre, propionate has the highest affinity for FFAR 2. Furthermore, propionate is an end product of bacterial metabolism, and thus, unlike acetate, does not undergo conversion to other SCFAs. Increasing colonic propionate is therefore an attractive target for appetite modulation.

We have developed a novel delivery system for delivering propionate to the right site in the colon and we now wish to optimise the delivery of propionate to the colon in man using stable isotope labelling methods.

DETAILED DESCRIPTION:
The role of SCFA in appetite regulation: SCFA have been shown to stimulate PYY and GLP-1 production in animal models and dietary fibre, of which SCFA are the major end products, induce appetite regulation in humans. However the evidence underpinning which dietary fibres induce appetite regulation in humans is very weak because of the difficulty in controlling studies with very high fibre intake. In a recent project funded under the BBSRC DRINC initiative (BB/H004815/1), we have the first direct evidence that SCFA can directly regulate appetite in humans. Prior to this study, in order to achieve production of SCFA to a level, which is high enough to induce appetite-regulating effects, very large amounts of dietary fibre (>25 g/d and up to 40 g/d) are required, and compliance with high fibre diets is poor due to gastrointestinal side effects. Furthermore, supplementing diets with mixed high fibre does not predictably or reliably increase colonic SCFA production or circulating levels of SCFA in all human populations because of the variability in gut microbial activity. Finally, orally administered SCFAs are not palatable and are rapidly absorbed in the small intestine where L cells are sparse. In our studies to date we have focussed on the SCFA propionate because it has the highest affinity for the receptors and is an end product of metabolism in the microbiota and therefore seems the obvious target to manipulate to investigate the effects of SCFA on appetite regulation. To overcome the unpalatably high levels of fermentable dietary fibre needed to significantly increase colonic propionate levels, and the unpredictability in the production of the resulting SCFAs, we have developed and tested a novel delivery system targeting the release of gram quantities of propionate in the proximal colon. We estimate that our delivery system may lead to a 2-8 fold increase in colonic propionate, a level very difficult to achieve through feeding a mixed fermentable fibre diet. This level of propionate production might have been observed in ancestral diets and in parts of rural Africa where dietary fibre intake is very high. We have also demonstrated that delivery system increases plasma propionate levels, reduces food intake in acute studies of appetite, and in a longer term study (24 weeks), positive effects on food intake, body composition, glucose homeostasis, circulating lipids, cholesterol and liver function, liver and visceral fat and weight management were observed. However, in these studies we pragmatically chose an preparation that could be produced at scale. The amount of propionate released can be varied which in itself may affect the rate and amount of propionate released. For an ingredient, with the potential to be incorporated into a wide variety of foodstuffs, we now wish to investigate the optimum delivery system preparation that delivers the maximal propionate dose in the least amount of material.

We plan to use non-invasive, stable isotope labelling methodologies to determine propionate bioavailability from a range of delivery system preparations, in order to determine the optimum preparation for delivering maximal propionate to the proximal colon.

ELIGIBILITY:
Inclusion Criteria:

* overweight males (BMI 25-35 kg/m2) aged between 21 - 65

Exclusion Criteria:

* Weight change of > 3kg in the preceding 2 months
* Current smokers
* Substance abuse
* Excess alcohol intake
* Pregnancy
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease
* Kidney disease
* Liver disease
* Pancreatitis
* Use of any medication

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to maximal 13C appearance in breath | over 24 hrs
  The time to peak maximal excretion in breath 13C (measured in breath 13CO2) will be the primary outcome criterion

SECONDARY OUTCOMES:
Area under curve of breath 13C excretion | over 24hrs
  The area under the curve of breath 13C excretion (measured in 13CO2) will be determined to assess amount of propionate released.

OTHER OUTCOMES:
Effect of preparations on appetite | 0ver 8 hrs
  The effect of different delivery system preparations on appetite will be determined by visual analog scale measurements and ad libitum food intake

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Morrison, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Glasgow Clinical Research Facility, Glasgow, Lanarkshire, United Kingdom